CLINICAL TRIAL: NCT03291223
Title: Gaucher Disease Outcome Survey (GOS)
Status: Recruiting | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: GOS
Record Dates: First submitted 2017-08-08; First posted 2017-09-25 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GOS Participants: GOS is a disease specific registry open to all Gaucher patients irrespective of treatment status or type of treatment

SUMMARY:
The Gaucher Outcomes Survey (GOS) is an ongoing observational, international, multi-center, long-term Registry of Patients with Gaucher Disease irrespective of their treatment status or type of treatment received. No experimental intervention is involved. Patients undergo clinical assessments and receive care as determined by the patients' treating physician.

The objectives of the registry include to evaluate the safety and long-term effectiveness of velaglucerase alfa, to characterize patients receiving velaglucerase alfa or other Gaucher Disease-specific treatments, to gain a better understanding of the natural history of GD and to serve as a database for evidence-based management of Gaucher Disease over time in real-life clinical practice.

DETAILED DESCRIPTION:
20 MAY 2020: The temporary enrollment stop of new patients into this study due to the COVID-10 pandemic has been lifted in one or more countries/sites, and the study is now again enrolling new patients. However, some countries/sites may still have paused the enrollment of new patients due to the pandemic.

24 APRIL 2020: Enrollment of new patients into this study has been paused due to the COVID-19 situation. The duration of this pause is dependent on the leveling and control of the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age or gender with confirmed diagnosis (biochemical and/or genetic) of Gaucher disease
* Signed and dated written informed consent from the patient or, for patients aged <18 years (<16 years in the United Kingdom [UK]), their parent and/or legally authorized representatives (LAR), and assent of the minor where applicable. Legally authorized representatives are also applicable for cognitively impaired patients.

Exclusion Criteria:

- Patients currently enrolled in ongoing blinded clinical trials (drugs or devices; includes all blinded trials)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: GOS is a disease specific registry irrespective of treatment or treatment status, open to all patients of any age or sex with Gaucher disease of any type. Patients included may be those who are untreated, naive to therapy, individuals who are currently or have been previously treated with velaglucerase alfa (VPRIV), or individuals who have been receiving or are currently exposed to other treatments for Gaucher disease. There is no predefined sample size.
Sampling Method: Non-Probability Sample
Enrollment: 1257 (Estimated)
Dates: Start 2010-07-27 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline to one year for up to 20 years
  Treatment-emergent adverse events (TEAEs) are defined as adverse events (AEs) that either commenced or worsened following the first dose of VPRIV.
Number of Participants With Infusion-related Reactions (IRRs) | Baseline to one year for up to 20 years
  An IRR is defined as an AE that has been assessed as at least possibly related to treatment with VPRIV and occurs during an infusion or up to 24 hours post-VPRIV infusion.
Increase of Hemoglobin Concentration | Baseline to one year for up to 20 years
  Hemoglobin concentration will be assessed.
Increase of Platelet Count | Baseline to one year for up to 20 years
  Platelet count will be assessed.
Decrease in Liver Volume | Baseline to one year for up to 20 years
  Liver volume will be assessed by abdominal imaging.
Decrease in Spleen Volume | Baseline to one year for up to 20 years
  Spleen volume will be assessed by abdominal imaging.
Increase in Bone Mineral Density (BMD) | Baseline to one year for up to 20 years
  Bone mineral density will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Shire Study Physician, Study Director — Shire
Locations (1):
- Central Contact, Lexington, Massachusetts, United States

REFERENCES:
- [Derived] Ain NU, Vaishnaw M, Mistry PK. Natural-History Mapping of Lysosomal Storage Disorders (LSDs): Gaucher Disease as a Model for Precision Care. J Inherit Metab Dis. 2026 Jan;49(1):e70128. doi: 10.1002/jimd.70128. PMID 41527340
- [Derived] Revel-Vilk S, Ramaswami U, Pintos-Morell G, Hughes D, Nicholls K, Reisin R, Giugliani R, Goker-Alpan O, Istaiti M, Gill A, Scarpa M, Botha J. Safety analysis of self-administered enzyme replacement therapy using data from the Fabry Outcome and Gaucher Outcome Surveys. Orphanet J Rare Dis. 2025 Mar 28;20(1):145. doi: 10.1186/s13023-024-03416-2. PMID 40155993
- [Derived] Elstein D, Belmatoug N, Bembi B, Deegan P, Fernandez-Sasso D, Giraldo P, Goker-Alpan O, Hughes D, Lau H, Lukina E, Revel-Vilk S, Schwartz IVD, Istaiti M, Botha J, Gadir N, Schenk J, Zimran A; GOS Study Group. Twelve Years of the Gaucher Outcomes Survey (GOS): Insights, Achievements, and Lessons Learned from a Global Patient Registry. J Clin Med. 2024 Jun 19;13(12):3588. doi: 10.3390/jcm13123588. PMID 38930117
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fcd4db2bf003ab4662b